CLINICAL TRIAL: NCT04370730
Title: Dimensional and Developmental Approach to Psychotic Episodes in Children and Adolescents: Impact on Clinical Management
Brief Title: Dimensional and Developmental Profiles of Psychosis in Children and Adolescents
Acronym: PSYDEV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K160906J; 2018-A01072-53 (Other: ANSM)
Record Dates: First submitted 2020-03-25; First posted 2020-05-01 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-01

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: schizophrenia; schizophrenia spectrum; psychosis; early-onset; cognition; magnetic resonance imaging; course of illness; treatment response
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Disease Progression | interventions — Neuroimaging

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prospective cohort (Other): prospective monitoring of children and adolescents with schizophrenia and related psychotic disorders
  Interventions: Other: clinical, neuroimaging and DNA assessments

INTERVENTIONS:
Other: clinical, neuroimaging and DNA assessments — Selected assessments, including evaluation of treatment response to specific antipsychotic drugs, will be performed at follow-up visits after 1, 3 and 5 years

SUMMARY:
Five collaborating sites in France will study the broad spectrum of schizophrenia in children and adolescents. Patients will be studied with diagnostic interviews, developmental histories, dimensional clinical ratings, comprehensive cognitive assessments, neuroimaging and DNA (copy number variant) analyses (in families and patients who agree), and follow-up of course of illness, cognitive status and treatment response to specific antipsychotic drugs. The goal of the study is to test a prior hypothesis about clinical subgroups in this population and to test whether these subgroups predict antipsychotic medication response.

DETAILED DESCRIPTION:
This study relates to the organization of a collection of clinical, biological / genetic and radiological (MRI) data from people with a psychotic episode and from their families. These data will be analyzed to clarify whether there is a different response to antipsychotic treatment based on developmental and clinical expression.To answer the question asked in the research, it is planned to include people with at least one psychotic episode,The target population will be a prospective cohort of patients admitted to a hospital or psychiatric clinic for the treatment of psychotic symptoms.Comprehensive medical evaluation will be carried out according to the clinical features and medical history of each patient, to identify medical causes of psychosis. Comprehensive neuropsychological and speech / language evaluation will be completed. A child psychiatrist-diagnostician will complete the Lifetime Dimensions of Psychosis Scale - Child and Adolescent version at baseline. When the patient and parents agree, structural and functional MRI examinations will also be completed, and blood will be drawn for DNA extraction and analysis. Selected assessments (including evaluation of treatment response to specific antipsychotic drugs) will be performed at follow-up visits after 1, 3 and 5 years.

ELIGIBILITY:
Inclusion Criteria for the Patient:

1. Children and young adults ages 7-20 years with age of onset of psychotic disorder between 7-17 years.
2. Hospitalized or seen for out-patient treatment for a psychotic episode, acute or chronic.
3. DSM-V diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, brief psychotic disorder, psychotic disorder not otherwise specified, or major depressive episode with psychotic features.
4. Written informed consent signed by the parents or the individual(s) with legal parental authority, and by the minor patient if his/her condition permits.
5. Written informed consent signed by the patient if he/she is a major, after clinical stabilization (not delusional).
6. Has health insurance coverage from Social Security (France) (not AME coverage).

Inclusion Criteria for parents or siblings wishing to participate in the genetic part of the study :

1. Parents : no specific criteria.
2. Siblings : siblings are eligible to participate if there are at least two first-degree relatives with psychotic disorders (including the patient) in the family.
3. Written informed consent for the genetic part of the study signed by any participating parents and siblings.
4. Has health insurance coverage from Social Security (France) (not AME coverage).

Exclusion Criteria:

1. Moderate or severe intellectual deficiency (IQ < 50).
2. Psychoses judged to be secondary to medical illness, medication effects or drugs of abuse.
3. Diagnosis of bipolar disorder.
4. Patients who are under legal guardianship.
5. For the neuroimaging part of the study only : any contraindications to Magnetic Resonance Imaging.

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Lifetime Dimensions of Psychosis Scale-Child and Adolescent Version | 4 months
  Symptoms are rated for lifetime duration and for severity during the worst two-week period.
  Number of participants assigned to each of four clinical clusters derived by cluster analysis from clinical and developmental ratings on this scale as previously described.

SECONDARY OUTCOMES:
Clinical global impressions scale - change version | at 5 years
  score on a 7 point scale ; worse is 7
Cortical gray matter volume (Magnetic Resonance Imaging) | up to 4 months
  Statistical differences among the four clinical clusters in the summary measure of cortical gray matter volume
Stability of clinical profile on Lifetime Dimensions of Psychosis Scale-Child and Adolescent Version | at 5 years
  differences among the four clinical clusters over time, comparing the cluster assignment at the time of stabilization to the assignment at the last study visit

CONTACTS AND LOCATIONS:
Overall Officials: Claudine LAURENT-LEVINSON, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (6):
- France (6):
  - Fondation Vallée, Gentilly, Gentilly
  - CHRU de Lille, Lille
  - CHU de Nice, Nice
  - Pitié Salpétrière, Paris
  - CHU de Rouen, Rouen
  - CHU de Rouvray, Rouen

IPD SHARING:
Plan to Share IPD: Undecided